CLINICAL TRIAL: NCT04234048
Title: A Phase 1a/1b Trial in Relapsed/Refractory T-cell Non-Hodgkin Lymphoma to Determine the Safety Profile, Pharmacology, and Maximum Tolerated Dose of ST-001, a Fenretinide Phospholipid Suspension (12.5 mg/mL) for Intravenous Infusion
Brief Title: Phase 1 Trial of ST-001 nanoFenretinide in Relapsed/Refractory T-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SciTech Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-001-010
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: T-cell Lymphoma; Cutaneous/Peripheral T-Cell Lymphoma; Peripheral T-cell Lymphoma; Peripheral T-Cell Lymphoma, Not Classified; Primary Cutaneous T-cell Lymphoma; Cutaneous T-Cell Lymphoma, Unspecified; Cutaneous T-cell Lymphoma; Follicular T-Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Sézary's Disease; Mycosis Fungoides
Keywords: Lymphoma; CTCL; Sézary syndrome; mycosis fungoides; PTCL; AITL; cALCL
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Immunoblastic Lymphadenopathy; Sezary Syndrome; Mycosis Fungoides; Lymphoma | interventions — Fenretinide; MAC-ST-001

STUDY DESIGN:
Intervention Model Description: Dose escalation oncology Phase 1 with extended cohort study (1b); Up to 46 patients for the whole study: up to 8 patients for accelerated phase 1a (single patient cohort) + up to 18 patients for standard phase 1a (3+3 design) + 20 patients for phase 1b at the maximum tolerated dose (MTD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 (Experimental): Accelerated Phase 1a + Standard Phase 1a + Phase 1b
  Accelerated Phase 1a
  Up to 9 patients for accelerated phase 1a (single patient cohort); dose levels of ST-001 nanoFenretinide (mg/m^2/day X 5 days every 21 days):
  Dose Level 1 1.25 (1 patient) Dose Level 2 2.5 (1 patient) Dose Level 3 5.0 (1 patient) Dose Level 4 10 (1 patient) Dose Level 5 20 (1 patient) Dose Level 6 40 (1 patient) Dose Level 7 80 (1 patient) Dose Level 8 160 (1 patient) Dose Level 9 320 (1 patient)
  Standard Phase 1a
  Up to 15 patients for standard phase 1a (3+3 design); dose level (mg/m2/day X 5 days every 21 days):
  Dose Level 10 640 (3-6 patients) Dose Level 11 896 (3-6 patients) Dose Level 12 1,254 (3-6 patients) Dose Level 13 1,756 (3-6 patients)
  Phase 1b
  20 patients for phase 1b at the maximum tolerated dose (MTD)
  Interventions: Drug: Fenretinide

INTERVENTIONS:
Drug: Fenretinide — Accelerated Phase 1a 100% Dose escalation in 8 single-patient cohorts
  Standard Phase 1a 40% Dose escalation in 3-patient cohorts X 3 cohorts
  Phase 1b Dosed at MTD in 20 patients as disease-specific expanded cohort
  Other Names: nanoFenretinide; ST-001; 4-HPR; N-(4-hydroxyphenyl)retinamide; N-(4-hydroxyphenyl)-all-trans-retinamide

SUMMARY:
This study evaluates a fenretinide phospholipid suspension for the treatment of T-cell non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Fenretinide has been shown to be a relatively safe and effective anticancer therapy; however, dose limiting toxicities due to the excipients used in previous formulations has impeded its therapeutic utility. The product formulation in the current study (ST-001) is a phospholipid suspension of nanoparticle sized fenretinide. The current study is a Phase 1 trial in relapsed/refractory (R/R) T-cell non-Hodgkin's lymphoma in order to determine the safety profile, pharmacology, and maximum tolerated dose (MTD) of ST-001 nanoFenretinide. Targeted T-cell non-Hodgkin's lymphoma (T-Cell NHL) indications include: (1) Cutaneous T-cell lymphoma (CTCL) including mycosis fungoides (MF) and Sézary Syndrome (SS); (2) non-cutaneous T-cell lymphoma (non-CTCL) subtypes: angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma (PTCL) not otherwise specified (NOS); and, follicular T-cell lymphoma (FTCL) as defined in the 2016 revision of the WHO classification of lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed diagnosis of the following specific types of T-cell lymphomas (TCL):

  1. Cutaneous T-cell lymphoma (CTCL): mycosis fungoides (MF), Sézary Syndrome (SS), or primary cutaneous CD30+ anaplastic large cell lymphoma (cALCL).
  2. Nodal TCL: Peripheral T-cell lymphoma (PTCL) not otherwise specified (NOS), angioimmunoblastic T-cell lymphoma (AITL), or follicular T-cell lymphoma (FTCL) as defined in the 2016 revision of the WHO classification of lymphoid malignancies[98] (Appendix A).
* For standard phase 1a and expanded cohort (1b): Patients must all have at least one measurable disease site using criteria provided in section 11.
* Relapsed or refractory (R/R) disease, after at least 1 prior treatment regimen as per disease staging (including but not limited to oral bexarotene, interferon, any oral or IV HDAC inhibitor, any topical, oral or IV chemotherapy drugs, radiotherapy, retinoids, topical steroids, systemic steroids, phototherapy, immunomodulators, Biologics and others based on PI discretion. Refer to section 2.1 of the protocol for more details).
* Refractory disease is defined as lack of objective response (i.e., partial or complete response) to most recent therapy.
* Relapsed disease is defined as recurrent disease after prior therapy that does not qualify as refractory disease.
* Other systemic treatments not specified may be allowed based on PI judgement in consultation with the Sponsor.
* For primary cutaneous lymphomas, stage IB, II, III and IV according to the TNMB system (Appendix C) are eligible. For primary nodal lymphomas, patients with stages II-IV according to the Ann Arbor staging system are eligible.
* Minimum of 4 weeks must have elapsed since last systemic treatment or radiation therapy treatment (or 6 weeks for any nitrosourea-containing regimens), and patients must have recovered from all toxicity of last treatment. If the PI assesses that it is in the best interest of the patient to have a shorter washout period, they may submit a written request to the sponsor and can enroll the patient after written approval has been received.
* Age ≥18 years. Both genders are included. However, women of childbearing potential must have a negative B-HCG serum pregnancy test (see Section 10 Study Calendar, Pre-Study, footnote b) and agree to use effective contraceptive methods for the duration of the study. A urine pregnancy test is required just prior to the first dosing session of every treatment cycle.
* ECOG performance status 0-1 (Karnofsky ≥60%, see Appendix B).
* Life expectancy greater than 6 months.
* Patients must have normal organ and marrow function as defined below:
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin within normal institutional limits. Patients with total bilirubin ≤ 1.5 X upper limit of normal are eligible
* AST (SGOT) and ALT (SGPT) within institutional upper limit of normal
* Creatinine clearance ≥60 mL/min/1.73m2 by the Modification of Diet in Renal Disease (MDRD) equation

Or if the patient were to have bone marrow involved NHL, the hematological requirements should be as listed below:

* Absolute neutrophil count ≥ 500/μL
* Platelets ≥ 50,000/μL
* Triglyceride blood level (fasting) <300mg/dL at time of enrollment (normal: <150mg/dL; borderline high = 150-199mg/dL; high = 200-499mg/dL; very high = 500mg/dL or higher).
* ST-001 is an experimental drug and the risks to the unborn or nursing child are unknown. Pregnant or breastfeeding women cannot take part in this study. Women of childbearing age are required to have a blood and/or urine pregnancy test before beginning the investigational study treatment. If you are sexually active, it is important that you not become pregnant or father a child because this medication may be harmful to your unborn child. Patients must discuss pregnancy plans with their doctor before enrolling in this study and agree that they will take the appropriate precautions not to become pregnant while enrolled in the study.

If there is any chance that patient can get pregnant, patient must either agree to not have vaginal intercourse or you must use two (2) types of birth control (hormonal, barrier method of birth control, abstinence) at the same time. These birth control methods must be used from the time of enrollment, all during investigational study treatment including during temporary breaks from therapy, and for at least 4 months after the last dose of ST-001.

• Informed consent of the patient or a legal authorized representative (LAR) must be obtained prior to any study related procedures.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known or history of central nervous system (CNS) disease are excluded from this clinical trial because of their poor prognosis and because of concerns regarding toxicity attribution.
* History of allergic reactions or sensitivity to retinoids or to any excipients of ST-001.
* Concomitant drug administration.

Patients who require concurrent treatment with drugs that are strong CYP3A inducers are excluded from the trial. Patients who have been treated previously with strong CYP3A inducers may enroll in the trial and receive their first dose of ST-001 only after four weeks have elapsed since the last dose of the CYP3A inducer. Strong inducers of human CYP3A include barbiturates, bosentan, carbamazepine, efavirenz, enzalutamide, etravirine, systemic glucocorticoids, mitotane, modafinil, nevirapine, oxcarbazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, troglitazone as well as the OTC herbal product St John's Wort (https://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm#table2-3; http://www.mayomedicallaboratories.com/it-mmfiles/Cytochrome_P450_3A4_and_3A5_Known_Drug_Interaction_Chart.pdf; http://oncologypro.esmo.org/content/download/66542/1203090/file/CYP3A-inhibitors-inducers-DDI.pdf)

Patients who require concurrent treatment with drugs that are strong to moderate CYP3A inhibitors are excluded from the trial, and patients who have been treated previously with strong CYP3A inhibitors may enroll in the trial and receive their first dose of ST-001 only after four weeks have elapsed since the last dose of the CYP3A inhibitor. This group of inhibitors includes certain antivirals (boceprevir, danoprevir, paritaprevir; elvitegravir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, telaprevir, tipranavir; ombitasvir, dasabuvir), macrolide antibiotics (e.g., clarithromycin, erythromycin, telithromycin, troleandomycin) and ciprofloxacin, antifungals (e.g., clotrimazole, fluconazole, ketoconazole, itraconazole, nefazodone, posaconazole, voriconazole), aprepitant, cimetidine, cobicistat, conivaptan, crizotinib, cyclosporine, diltiazem, dronedarone, idelalisib, luvoxamine, imatinib, tofisopam, suboxone and verapamil as well as dietary grapefruit juice and grapefruit (https://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm#table2-3; http://www.mayomedicallaboratories.com/it-mmfiles/Cytochrome_P450_3A4_and_3A5_Known_Drug_Interaction_Chart.pdf; http://oncologypro.esmo.org/content/download/66542/1203090/file/CYP3A-inhibitors-inducers-DDI.pdf)

If patients being treated with ST-001 require the use of drugs that are either strong inducers of CYP3A or strong to moderate inhibitors of CYP3A to treat a medical condition, all treatment with ST-001 should be discontinued immediately and no further treatment with ST-001 will be allowed.

Use of acetaminophen, cephalosporins and other known hepatotoxic agents is allowed with caution and close monitoring, due to known or potential interaction with ST-001 and potential increased risk of hepatotoxicity[52]. Patients who require replacement therapy with oral steroids should be allowed to continue the treatment if treatment with stable dose has been initiated more than 2 weeks prior to beginning ST-001 infusion. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/. Medical reference texts such as the Physicians' Desk Reference may also provide this information.

As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Physician investigators should consult the websites listed above for the most current information regarding drug interactions via CYP3A isozymes.

Use of vitamin A supplements is prohibited. Standard multivitamin doses are allowed.

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NY heart classification III/IV), unstable angina pectoris, cardiac arrhythmia, QTc interval >450 milliseconds on baseline triplicate ECG, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ST-001is a retinoid agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ST-001, breastfeeding should be discontinued if the mother is treated with ST-001.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ST-001. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with any active hepatitis infections.
* Presence of nyctalopia (night blindness), or hemeralopia (defective vision in a bright light, 'day blindness') at enrollment, or any other retinal, ophthalmological condition (eg: retinitis pigmentosa, choroidoretinitis and xerophthalmia), and glaucoma.
* Patients who have received prior fenretinide systemic therapy
* Patients with T-cell lymphoma types other than those specified in section 3.1.1 are not eligible even if they have cutaneous dissemination. Similarly, patients with any type of natural killer (NK)- or B-cell lymphoma are not eligible regardless of sites of involvement by disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 12 months
  To determine the MTD of ST-001 nanoFenretinide (12.5mg/mL) for IV infusion in patients with CTCL and other T-cell NHL.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 12 months
  The number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0 will be determined. All patients who receive any dose of ST-001 will be evaluable for toxicity. The incidence rates of adverse events (AEs) will be tabulated by system organ class and preferred term, and by severity. All AEs with corresponding attributes will be displayed in a by-patient listing. The investigator at each site will determine the causal relationship between study medication and AEs. Subsets of AEs to be summarized include Severe Adverse Events (SAEs), suspected treatment-related AEs, and AEs that resulted in withdrawal of treatment or death.
Number of participants with complete response (CR) or partial response (PR) to ST-001 | 24 months
  Any patient who has at least one measurable disease site and has received at least on full cycle (5-day infusion) of ST-001 is eligible for response-to-treatment evaluation. The frequency and proportion of subjects with CR or PR will be calculated with a 95% Clopper Pearson confidence interval. CR + PR will constitute the overall response rate (ORR). The Global Response Scale (GRS) will be used to determine response of CTCL patients to ST-001. The GRS incorporates all components of the TNMB system (skin, lymph nodes, viscera, and blood). The International Working Group (IWG) Criteria for Response Assessment will be used to determine response in non-CTCL T-NHL patients.
Fenretinide Cp(plateau), half-life (t1/2), and calculated parameters of Clearance and Volume of Distribution | 18 months
  Pharmacokinetic (PK) evaluation of fenretinide Cp X t curves, Cp(plateau), and half-life (t1/2) as well as calculated parameters of Clearance and Volume of Distribution will be conducted at each dose level when all of its planned first cycle treatments have been completed. PK analysis will use descriptive statistics to characterize the range, median, and mean of calculated values of fenretinide clearance, volume of distribution, and distribution and elimination phase half-lives across all evaluable patients using individual patient C X t data. The relationship between dose and CpMAX and/or AUC will be examined as will their relationship to grade of toxicity.
Activation of cytolytic T-lymphocytes (CTLs) and natural killer (NK) cells after ST-001 treatment. | 24 months
  The pharmcodynamic (PD) effect of ST-001 will be evaluated in tissue biopsies taken from tumorous skin lesions of CTCL patients. CTL and NK cell activation will be measured by expression of granzyme A and B, perforin, and NKG2D using immunohistochemical staining (IHC) of tissue biopsies. In addition, CTLs and NK cell tumor infiltration will be evaluated using CD8 and CD56 IHC staining, respectively. Biomarker analysis will use each patient's baseline (pre-treatment) values as the Control value and normalize PD changes as % change from baseline. In addition, the baseline PD biomarker values across all evaluable patients will be characterized as a distribution, and the on-treatment PD responses analyzed for values that are statistical outliers from the baseline distribution of values.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Moiin, MD, Study Director — SciTech Development, Inc.; Oleg E Akilov, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center (UPMC); Ann F Mohrbacher, MD, Principal Investigator — University of Southern California; Barbara Pro, MD, Principal Investigator — Columbia University; Dipenkumar Modi, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Auris O Huen, MD, PharmD, Principal Investigator — M.D. Anderson Cancer Center; Ryan A Wilcox, MD, PhD, Principal Investigator — University of Michigan; Brad Haverkos, M.D., Principal Investigator — University of Colorado, Denver; Christiane Querfeld, M.D., Ph.D., Principal Investigator — City of Hope Medical Foundation; Aaron R Mangold, M.D., Principal Investigator — Mayo Clinic; Jonathan Moreira, M.D., Study Director — Northwestern University, Robert H. Lurie Comprehensive Cancer Center
Locations (10):
- United States (10):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope Medical Foundation, Duarte, California
  - University of Southern California, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No